CLINICAL TRIAL: NCT01289808
Title: Reduced Infant Response To A Routine Care Procedure After Glucose 25% Analgesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: changes were made to the which needed an entireley new submission
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Shay Barak, Senior Neonatologist, The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SAOR 005.CTIL
Record Dates: First submitted 2011-01-27; First posted 2011-02-04 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Infant; Newborn Diseases
Keywords: Glucose; analgesic; newborns
MeSH Terms: interventions — Water; Injections

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- glucose 25% (Experimental): 180 healthy babies born term in the Baruch Padeh Medical Center, Poriya.
  There will be three study groups:
  Study Group: 60 newborn infants who will receive 1cc 25% Glucose, 2-3 minutes prior red-reflex examination.
  Base line (control) Group 1: 60 newborn infants who will receive 1cc Water for Injection (WFI), 2-3 minutes prior red-reflex examination.
  Base line (control ) Group 2: 60 newborn infants who will not receive neither glucose nor Water for Injection (WFI), 2-3 minutes prior red-reflex examination
  Interventions: Drug: Glucose 25%

INTERVENTIONS:
Drug: Glucose 25% — 1ml of glucose 25% once
  Other Names: Water for injection
Drug: Glucose 25% — 1ml glucose once per os
  Other Names: water for injection once per os

SUMMARY:
Glucose has analgesic and calming effects in newborns. To date, it is not known whether the beneficial effects extend to care giving procedures that are performed after painful procedures. The investigators objective is to determine the effect of glucose 25% analgesia for procedural pain on infant pain responses during a subsequent care giving procedure.

DETAILED DESCRIPTION:
Pain in the newborn and young infant is a source of stress for the infant, family and care providers.

During hospitalization, a neonate undergoes a number of necessary procedures that may be either painful or cause discomfort to the baby.

Pain experienced during the neonatal period is known to have long term effects on the baby.

The red-reflex test is a routine examination performed on a neonate after birth and once again before discharge from the hospital. The examination causes discomfort to the infant.

Glucose has analgesic and calming effects in newborns. To date, it is not known whether the beneficial effects extend to care giving procedures that are performed after painful procedures. Our objective is to determine the effect of glucose 25% analgesia for procedural pain on infant pain responses during a subsequent care giving procedure.

ELIGIBILITY:
Inclusion Criteria:

* Full term above 37 weeks gestation.
* Normal birth-weight, healthy infants
* Males and Females
* Whose parents have signed the informed consent form

Exclusion Criteria:

* Premature born below 37 weeks
* Chromosomal abnormalities or congenital malformation.
* Suffering neurological imbalance
* Inability of oral feeding

Ages: 1 Day to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Reduced infant response to a routine care procedure after glucose 25% analgesia | 30 minutes
  An observer nurse will focus on the infant's facial expression. A score between 0 and 3 will be assigned for each of the three facial expression indicators.
  For physiological data, infants will be monitored for changes in heart rate and oxygen saturation using a transcutaneous pulse oximeter. A score between 0 and 3 will be assigned for each of the physiological indicators

CONTACTS AND LOCATIONS:
Overall Officials: Shay Barak, MD, Principal Investigator — Neonatal Department, The Baruch Padeh Medical center - Poria